CLINICAL TRIAL: NCT06874673
Title: A Multicenter, Prospective, Double-Blind Randomized Controlled Trial Evaluating the Efficacy and Safety of Pronase in Improving Endoscopic Mucosal Clarity During Colonoscopy for Patients with Colitis
Brief Title: Pronase in Improving Endoscopic Mucosal Clarity During Colonoscopy for Patients with Colitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Affiliated Hospital of Jiangnan University (Other); The Affiliated People's Hospital of Ningbo University (Other Government); Shanghai 8th People's Hospital (Other); Huashan Hospital (Other); Shanghai Baoshan District Wusong Central Hospital (Unknown); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Pudong Hospital (Other); The People's Hospital of Leshan (Other); Shanghai Pudong New Area Gongli Hospital (Other); Huadong Hospital (Other); Shanghai Songjiang District Central Hospital (Unknown); Jinshan Hospital Fudan University (Other); Dongfang Hospital Affiliated to Tongji University (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept and Digestive Endoscopy Center, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CHEC2024-330
Record Dates: First submitted 2025-03-05; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pronase; Mucosal Clarity
Keywords: Pronase; Colonoscopy; Mucosal Clarity; Colitis; Ulcerative Colitis; Crohn's Disease; inflammatory bowel disease
MeSH Terms: conditions — Colitis; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Pronase; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pronase Group (Group A) (Experimental): During colonoscopy, the mucosal surface of the intestine was rinsed with a pronase solution to remove mucus.
  Interventions: Drug: Pronase
- Saline Group (Group B) (Placebo Comparator): During colonoscopy, the mucosal surface of the intestine was rinsed with saline solution to remove mucus.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Pronase — During the colonoscopy procedure on participants in Group A, when colitis with mucosal mucus impeding visualization is encountered, the gastroenterologist uses a solution of pronase (200 U/mL) delivered through the endoscope's biopsy forceps to irrigate the affected area. Images are captured before and after the irrigation, and a score for improvement in mucosal clarity is assigned. The location of the lesion, irrigation time, and volume of fluid used are recorded. During endoscope withdrawal, the same area is reassessed for improvement in clarity, and the disease activity is evaluated. Biopsy specimens are taken from the most severe inflammation site for histopathological examination.
  Arms: Pronase Group (Group A)
Drug: Saline (NaCl 0,9 %) (placebo) — During the colonoscopy procedure on participants in Group B, when colitis with mucosal mucus impeding visualization is encountered, the gastroenterologist uses saline delivered through the endoscope's biopsy forceps to irrigate the affected area. Images are captured before and after the irrigation, and a score for improvement in mucosal clarity is assigned. The location of the lesion, irrigation time, and volume of fluid used are recorded. During endoscope withdrawal, the same area is reassessed for improvement in clarity, and the disease activity is evaluated. Biopsy specimens are taken from the most severe inflammation site for histopathological examination.
  Arms: Saline Group (Group B)

SUMMARY:
Pronase is a proteolytic enzyme known for its ability to clear mucus by breaking down its main component, mucin, through enzymatic hydrolysis. This property makes it useful in gastroscopy, where it is employed to improve the visibility of the mucosal surface during endoscopic examinations. Given the same mechanism, pronase may also be beneficial in enhancing mucosal clarity during colonoscopy. This multicenter, prospective, double-blind randomized controlled trial is designed to assess the effectiveness and safety of pronase in improving mucosal visibility in patients with colitis during endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with intestinal inflammation during colonoscopy, accompanied by mucus obscuring visualization, were included, particularly those with inflammatory bowel disease (IBD), regardless of the presence or absence of clinical symptoms such as abdominal pain, diarrhea, hematochezia, or mucoid stools.
* Researchers assessed the current health status of potential participants to ensure they could tolerate colonoscopy (based on physical examination and medical history).
* Age range was 18-75 years (inclusive).
* Participants provided written informed consent to participate voluntarily.

Exclusion Criteria:

* Participants with known hypersensitivity or allergy to the study medication.
* Participants with peritonitis, intestinal obstruction, severe intestinal infection, or radiation colitis.
* Participants who did not exhibit intestinal mucus obscuring endoscopic visualization during colonoscopy.
* Participants with severe cardiovascular, pulmonary, neurological, or renal disease, or those deemed unfit for colonoscopy.
* Participants who did not provide written informed consent or lacked the capacity to do so.
* Pregnant or breastfeeding women.
* Participants who had taken antiplatelet medications (e.g., aspirin, clopidogrel) or had abnormal coagulation function within 7 days prior to colonoscopy.
* Participants currently participating in other clinical observation trials or who had participated in another clinical trial within 60 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Improvement rate of intestinal mucosal clarity after rinsing | From the start of the rinse to 30 seconds after the end of the rinse.
  This is defined as a mucosal clarity improvement score of 3 or higher on colonoscopy after rinsing of the mucoid attachment site, signifying achievement of mucosal clarity improvement. The improvement rate is calculated as the percentage of participants within a group who achieve mucosal clarity improvement divided by the total number of participants in that group.

SECONDARY OUTCOMES:
Colonoscopist satisfaction score | From start to finish of the colonoscopy.
  This reflects the overall satisfaction of the colonoscopist with the effect of the rinsing solution on mucosal clarity, measured using a 5-point Likert scale.Scores range from 5 to 1, with higher scores meaning better results.
Rinsing solution volume | From the start of the rinse to 30 seconds after the end of the rinse.
  This is defined as the volume of liquid consumed during rinsing of the area with the most severe mucosal mucus adhesion in each case.
Ulcerative colitis endoscopic index of severity，UCEIS | From the start of the rinse to 30 seconds after the end of the rinse.
  The UCEIS score is a standardized tool for assessing the severity of inflammation in ulcerative colitis (UC) based on three core features: vascular Pattern, bleeding, and erosions/ulcers, as viewed through enteroscopy, with a total score of 0-8, with higher scores suggesting more severe lesions.
Endoscopic severity index of Crohn's disease, CDEIS | From the start of the rinse to 30 seconds after the end of the rinse.
  The CDEIS is based on the assessment of 4 parameters (deep ulcers, shallow ulcers, extent of surface involvement, and extent of ulcer involvement) in 5 sites (terminal ileum, right hemicolon, transverse colon, left hemisphere and sigmoid colon, and rectum), and the total score for an individual segment divided by the number of segments assessed, plus the presence or absence of stenosis yields a total score that ranges from 0 ~ 44 points, with higher scores suggestive of more severe lesions.
Simplified Geboes Score, SGS | From the start of the rinse to 30 seconds after the end of the rinse.
  The Simplified Geboes Score evaluates the degree of tissue inflammation by assessing neutrophils in the lamina propria, neutrophils in the epithelium and epithelial damage in the crypts and mucosal surfaces. The scale is as follows: grade 0 represents structural abnormalities or chronic infiltration without active inflammation; grade 1 represents basal plasmacytosis; grade 2 represents inflammatory cell infiltration in the lamina propria; grade 3 represents neutrophil infiltration in the epithelium; grade 4 represents crypt epithelial damage and grade 5 represents surface epithelial damage.
Colonic and ileal global histologic disease activity scores, CGHAS | From the start of the rinse to 30 seconds after the end of the rinse.
  The CGHAS scoring system evaluates mucosal inflammation levels in Crohn's disease patients through histological assessment of mucosal tissue biopsies. Its assessment parameters include: lamina propria inflammatory cell infiltration (e.g., neutrophils, mononuclear cells); chronic structural damage (e.g., crypt distortion, glandular architectural disarray); epithelial injury (e.g., erosions, ulcerations); and the extent of lesion involvement (quantified by the number of affected biopsy specimens). The scoring scale ranges from 0 to 16 points, with higher scores indicating more severe inflammatory activity.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-Shen Li, MD, PhD, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Naval Medical University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Kuo CH, Sheu BS, Kao AW, Wu CH, Chuang CH. A defoaming agent should be used with pronase premedication to improve visibility in upper gastrointestinal endoscopy. Endoscopy. 2002 Jul;34(7):531-4. doi: 10.1055/s-2002-33220. PMID 12170403
- [Background] Han JP, Hong SJ, Moon JH, Lee GH, Byun JM, Kim HJ, Choi HJ, Ko BM, Lee MS. Benefit of pronase in image quality during EUS. Gastrointest Endosc. 2011 Dec;74(6):1230-7. doi: 10.1016/j.gie.2011.07.044. Epub 2011 Oct 1. PMID 21963063